CLINICAL TRIAL: NCT01856348
Title: Effects of Vitamin D3 (1,25 Dihydroxyvitamin D3) on Pharmacokinetics and Absorption of Folic Acid and Fexofenadine in Healthy Volunteers
Brief Title: Vitamin D3, Folic Acid and Fexofenadine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PHA-11-VID/FOL-01
Record Dates: First submitted 2013-04-15; First posted 2013-05-17 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Physiological Effects of Vitamin D
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1, 25 dihydroxyvitamin D3 intake (Experimental): This is a single arm study.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D

SUMMARY:
The study is conducted to assess the effect of a vitamin D3 supplementation on the activities of two intestinal transporters and on the pharmacokinetics of the transporter substrates folic acid and fexofenadine.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

1. male or female
2. age 18 to 65 years at study entry
3. signed informed consent form
4. Body Mass Index > 18 - < 30 kg/m2
5. Participants must not have any other diseases (as assessed by the screening examination)
6. Participants must not take any concomitant medications except oral contraceptives in females
7. Normal blood count

Exclusion criteria:

1. Subjects with confirmed or suspected hypersensitivity towards the study medications
2. Contemporaneous participation in any other study
3. Females only: pregnancy
4. Females only: breast-feeding
5. Clinically significant abnormal laboratory findings
6. Known or suspected present or past malignancies of any kind
7. Known or suspected active infections, serious infections in the preceding 3 months
8. Positive hepatitis B, hepatitis C and / or HIV 1/2 serology
9. Subjects known or suspected not to comply with the study regulations
10. Subjects employed at the participating departments of the University Hospital Zürich.
11. Known or suspected present or past diseases which may interfere with the study
12. smokers
13. alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Ratio of the area under the concentration vs. time curve (AUC) of fexofenadine after vitamin D over AUC of fexofenadine before vitamin D | 10 days
  Changes in single-dose pharmacokinetics of racemic fexofenadine at the end of a substitution with 1,25 dihydroxyvitamin D3 in comparison to pharmacokinetics before the substitution.
Ratio of Area under the concentration vs. time curve (AUC) of folic acid after vitamin D over AUC of folic acid before vitamin D | 10 days
  Changes in single-dose pharmacokinetics of folic acid at the end of a substitution with 1,25 dihydroxyvitamin D3 in comparison to pharmacokinetics before the substitution.

SECONDARY OUTCOMES:
Number and characteristics of participants with adverse events | 10 days
transporter mRNA quantity | 10 days
  Comparison of transporter mRNA levels after ten days of vitamin D3 intake in comparison to the levels before intake.

CONTACTS AND LOCATIONS:
Overall Officials: Gerd A Kullak-Ublick, Prof MD, Principal Investigator — University Hospital Zurich, Pharmacology and Toxicology
Locations (1):
- University Hospital Zurich, Dept. of Clinical Pharmacology and Toxicology, Zurich, Canton of Zurich, Switzerland